CLINICAL TRIAL: NCT00227175
Title: Cornell Translational Behavioral Science Research Consortium: Hypertension Qualitative Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: N01-HC-25196 (0103-659); N01HC25196 (NIH)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
Keywords: African American; Hypertension; Medication adherence; Risk reduction
MeSH Terms: conditions — Hypertension; Medication Adherence; Risk Reduction Behavior

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Semi-structured, open ended interview

SUMMARY:
To explore the meaning, causes and treatment of hypertension in eligible patients. In addition the cultural, social, and psychological factors that either facilitate or serve, as barriers to behavioral change will be illuminated in this patient population.

DETAILED DESCRIPTION:
1. The first goal is to explore the meaning, causes and treatment of hypertension in eligible patients. In addition the cultural, social, and psychological factors that either facilitate or serve, as barriers to behavioral change will be illuminated in this patient population. Through a series of open-ended questions we will explore and build a better understanding of how hypertensive African American patients view their illness and the difficulties they have in taking their antihypertensive medications as prescribed.
2. The second goal of the qualitative phase is to use the responses obtained to inform how we should operationalize and tailor the positive affect induction and self-affirmation intervention methods in hypertensive African American patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be self-identified as African-Americans.
2. All patients must be aged 18 years and older.
3. All patients must be diagnosed as having hypertension: For this project, hypertension will be defined according to the widely accepted criteria of the 6th Joint National Committee (JNC VI) Guidelines on Prevention, Detection, Evaluation and Treatment of Hypertension, which is a systolic blood pressure > 140 mm hg or a diastolic blood pressure > 90 mm hg or if participants are taking any prescribed antihypertensive medication.
4. Patients must be able to provide informed consent in English.

Exclusion Criteria:

1. Patients who refuse to participate
2. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, MS, Principal Investigator — Weill Medical College of Cornell University; Gbenga Ogedegbe, MD, MS, Principal Investigator — Columbia University; Mary E Charlson, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

REFERENCES:
- [Background] Factors That Influence Medication Adherence Among African-Americans With Hypertension. Moore, JA, Boutin-Foster, C, Charlson, ME. Weill Medical College of Cornell University, New York, NY. Presented at the 12th Annual NHLBI Cardiovascular Minority Research Supplement Awardee Session, American Heart Association, November 2004.
- [Derived] Ogedegbe GO, Boutin-Foster C, Wells MT, Allegrante JP, Isen AM, Jobe JB, Charlson ME. A randomized controlled trial of positive-affect intervention and medication adherence in hypertensive African Americans. Arch Intern Med. 2012 Feb 27;172(4):322-6. doi: 10.1001/archinternmed.2011.1307. Epub 2012 Jan 23. PMID 22269592